CLINICAL TRIAL: NCT02478541
Title: Investigating Intra-hepatic Fatty Acid Partitioning and Its Regulation in Man. Studies to Understand the Role of Dietary Nutrients in Liver Fat Metabolism in Relation to Obesity in Man
Brief Title: Understanding Liver Fat Metabolism: Studies to Understand the Role of Dietary Sugars on Liver Fat Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Oxlip-2013_expt2
Record Dates: First submitted 2015-06-15; First posted 2015-06-23 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2016-11

CONDITIONS: Hypertriglyceridaemia
Keywords: triglycerides; glucose; fructose; fatty acids
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar Study_low fructose (Active Comparator): Consumption of a single test meal that contains fat and a sugary drink made with a low amount of fructose and high amount of glucose
  Interventions: Other: Sugar study
- Sugar Study_high fructose (Active Comparator): Consumption of a single test meal that contains fat and a sugary drink made with a high amount of fructose and low amount of glucose
  Interventions: Other: Sugar study

INTERVENTIONS:
Other: Sugar study — Subjects are given a single test meal on two study days that has a sugary drink that varies in the amount of fructose and glucose it contains. They consume the same amount of fat on both study days.

SUMMARY:
High levels of fatty substances in the blood increase the risk of developing coronary heart disease and having a heart attack. The investigators know a lot about one of these fatty substances, cholesterol. However, there is another fatty substance in the blood called triglyceride. The investigators do not understand much about what regulates the rate at which the liver produces triglyceride and liberates it into the bloodstream after eating a meal(s). The investigators are developing new techniques to measure these processes in healthy people. Ultimately a deeper understanding of the regulation of this process might lead to the development of new treatments for fat accumulation in the liver and high blood fat levels and related disorders. The present study is an investigation of how these processes relate to various bodily characteristics such as thinness and fatness and the distribution of fat in the body.

DETAILED DESCRIPTION:
The investigators will recruit men and women with no medical condition or relevant drug therapy that affects lipid, glucose or liver metabolism.

Purpose and design:

The investigators are asking the research question: "How does the amount and type of sugars consumed, such as those found in soft drinks, influence postprandial fatty acid and liver fat metabolism?"

It is known that consuming fructose by itself or with glucose can increase plasma triglyceride concentrations and liver fat amounts but it remains unclear how this happens.

To address this research question investigators want to undertake detail physiological studies, in a randomised cross-over study where individuals will be studied twice after the consumption of a single test meal that will contain different amounts of glucose and fructose with the same amount of dietary fat.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* BMI >19 <35kg/m2
* No medical condition or relevant drug therapy known to affect liver, lipid or glucose metabolism

Exclusion Criteria:

* Age <18 or >65 years
* Body mass index <19 or >35kg/m2
* A blood haemoglobin <120mg/dL
* Any metabolic condition or relevant drug therapy
* People who do not tolerate fructose
* Smoking
* History of alcoholism or a greater than recommended alcohol intake
* Pregnant or nursing mothers
* Women prescribed any contraceptive agent or device including oral contraceptives, hormone replacement therapy (HRT) or who have used these within the last 12 months
* History of severe claustrophobia
* Presence of metallic implants, pacemaker
* Haemorrhagic disorders
* Anticoagulant treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Plasma Triglycerides | 7 hours
  Postprandial plasma triglyceride concentrations will be measured biochemically, on a clinical analyser by taking regular blood samples from participants for a period of up to 7 hours after participants have consumed the test meal.

SECONDARY OUTCOMES:
Plasma glucose | 7 hours
  Postprandial plasma glucose concentrations will be measured biochemically, by taking blood samples from participants regularly after the consumption of a mixed test meal.

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Hodson, PhD, Principal Investigator — University of Oxford
Locations (1):
- Oxford Centre for Diabetes, Endocrinology and Metabolism, Oxford, United Kingdom